CLINICAL TRIAL: NCT03016702
Title: The Cognitive Resilience Study: Stress Tests for Alzheimer's Disease
Brief Title: The Cognitive Resilience Study
Acronym: CogRes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Bryan Alzheimer's Disease Research Center (Unknown); Duke University Center for the Study of Aging and Human Development (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Pro00078117; P30AG028716-11S1 (NIH); SPS # 224571 (Other: Duke University)
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2016-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Risk Alzheimer's Disease (Experimental): This group includes subjects with APOEe4 homozygotes, the genetic profile associated with the highest risk for late-onset AD and the next highest-risk group, APOE e3/e4 heterozygotes. To target the highest risk among the APOEe3/e4 heterozygotes in ADPR, the study team will consider TOMM40-'523 variant status. Although there is uncertainty about the independent role of TOMM40 in AD risk-stratification (especially across racial/ethnic groups), this study will use TOMM40-'523 to guide heterozygote selection based on findings that among e3/e4 heterozygotes, longer TOMM40-523 polyT sequences are associated with earlier age of onset for late-onset AD.
  Interventions: Other: Cognitive stress tests during functional MRI; Other: Cognitive stress tests during gait task
- Low Risk Alzheimer Disease (Experimental): This group includes e2/e2 homozygotes (rare) and e2/e3 heterozygotes. the genetic profile associated with low risk for late-onset development of Alzheimer's disease.
  Interventions: Other: Cognitive stress tests during functional MRI; Other: Cognitive stress tests during gait task

INTERVENTIONS:
Other: Cognitive stress tests during functional MRI — Subjects will undergo progressively more complex cognitive stress tests that assess memory and executive function while undergoing fMRI.
Other: Cognitive stress tests during gait task — Subjects will undergo progressively more complex cognitive stress tests that assess memory and executive function both in sitting and while ambulating on a force sensor mat.

SUMMARY:
The purpose of this study is to test whether two new cognitive "stress tests" may help distinguish between people at lower or higher genetic risk of Alzheimer's Disease. The investigators are trying to understand how these cognitive "stress tests" work in people who have not been diagnosed with Alzheimer's Disease and are not exhibiting symptoms of Alzheimer's Disease. Study subjects will undergo testing of memory and executive function during functional magnetic resonance image (fMRI) of the brain and also during a walking test.

DETAILED DESCRIPTION:
The objective is to establish the feasibility and evaluate the role of two novel tests of cognitive resilience for use in identification of early Alzheimer's Disease. The investigators hypothesize that exposure to the controlled stressor of increased cognitive task demand will evoke measurable phenotypes of poor resilience, which will be associated with Alzheimer's Disease risk. The study will include 30 volunteer participants from the Duke Alzheimer's Disease Prevention Registry (ADPR). The ADPR cohort has been characterized according to genetic risk based on genotype at loci associated with Alzheimer's Disease. The investigators will recruit a sample from the ADPR that includes 15 people in the "genetic high risk" group and 15 people, matched by age, in the "genetic low risk" group. Investigators and experimenters are masked to the genetic profile of all participants. All participants will undergo two cognitive stress test protocols. Both protocols include memory and executive function components, one done during functional MRI and one while ambulating on a force sensor mat. Both cognitive stress tests are minimal risk; the primary risk of this study is loss of confidentiality. Genetic testing is not performed as part of this protocol; the sampling strategy will make use of prior genetic testing results, which are not revealed to the primary investigators. In addition to determining whether scores on the two novel tests statistically differ by AD risk groups, the project will establish the tests' feasibility and characteristics for use in future study.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk 2 minutes without assistive device or assistance from another person
* Cognitive function within normal limits

Exclusion Criteria:

* Unable to undergo MRI
* Left handed
* Red/Green Color Blind
* Severe vision impairments
* Diagnosis of Alzheimer's Disease or other dementia/memory problem

Ages: 58 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Change in reaction time during memory testing during fMRI | Measured immediately during one hour fMRI
  The primary dependent variable will be change in reaction time when comparing a neutral memory task to a stress condition. Reaction time will be in ms and will be recorded while the subject is undergoing fMRI.
Change in reaction time during executive function testing during fMRI | Measured immediately during one hour fMRI
  The primary dependent variable will be change in reaction time when comparing a neutral executive function task to a stress condition. Reaction time will be in ms and will be recorded while the subject is undergoing fMRI.
Change in accuracy during memory testing during gait task | Measured immediately during one hour gait session
  The primary dependent variable will be DTEcog = (Dual task [cognitive score] - Single Task [cognitive score] / Single task [cognitive score]. For the memory task, the primary cognitive measure will be the number of correct responses.
Change in reaction time during executive function testing during gait task | Measured immediately during one hour gait session
  The primary dependent variable will be DTEcog = (Dual task [cognitive score] - Single Task [cognitive score] / Single task [cognitive score]. For the executive task, the primary cognitive measure in the DTEcog calculation will be reaction time.

SECONDARY OUTCOMES:
Change in accuracy during memory testing during fMRI | Measured immediately during one hour fMRI
  Secondary dependent variables are accuracy (% correct) when comparing a neutral memory task to a stress condition.
Change in accuracy during executive function testing during fMRI | Measured immediately during one hour fMRI
  Secondary dependent variables are accuracy (% correct) when comparing a neutral memory task to a stress condition.
Brain activation during memory testing during fMRI | Measured immediately during one hour fMRI
  Group differences in brain activation provoked by the memory stress condition will be assessed using brain maps that compare block-average BOLD signal for resting vs neutral task, resting vs stress task, neutral vs stress task.
Brain activation during executive function testing during fMRI | Measured immediately during one hour fMRI
  Group differences in brain activation provoked by the executive function stress condition will be assessed using brain maps that compare block-average BOLD signal for resting vs neutral task, resting vs stress task, neutral vs stress task.
Change in gait performance provoked by memory dual tasking | Measured immediately during one hour gait session
  The secondary dependent variable will be DTEmob = (Dual task[mobility score] - Single Task[mobility score] / Single task [mobility score]. For both memory and executive tasks, the mobility measure in the DTEmob calculation will be gait speed.
Change in gait performance provoked by executive function dual tasking | Measured immediately during one hour gait session
  The secondary dependent variable will be DTEmob = (Dual task[mobility score] - Single Task[mobility score] / Single task [mobility score]. For both memory and executive tasks, the mobility measure in the DTEmob calculation will be gait speed.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Whitson, MD, MHS, Principal Investigator — Duke University Aging Center
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No